CLINICAL TRIAL: NCT00458978
Title: Phase II Clinical Trial of AZD2171 Monotherapy in Recurrent or Metastatic Head and Neck Squamous Cell Carcinoma Patients
Brief Title: Cediranib Maleate in Treating Patients With Recurrent or Newly Diagnosed Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00148; NCI-2009-00148 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000538287; MGH-06-264; 06-264 (Other: Massachusetts General Hospital Cancer Center); 7309 (Other: CTEP); P30CA006516 (NIH); R21CA119591 (NIH)
Record Dates: First submitted 2007-04-09; First posted 2007-04-11 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Recurrent Hypopharyngeal Squamous Cell Carcinoma; Recurrent Laryngeal Squamous Cell Carcinoma; Recurrent Laryngeal Verrucous Carcinoma; Recurrent Lip and Oral Cavity Squamous Cell Carcinoma; Recurrent Metastatic Squamous Cell Carcinoma in the Neck With Occult Primary; Recurrent Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Recurrent Nasopharyngeal Keratinizing Squamous Cell Carcinoma; Recurrent Oral Cavity Verrucous Carcinoma; Recurrent Oropharyngeal Squamous Cell Carcinoma; Recurrent Salivary Gland Carcinoma; Salivary Gland Squamous Cell Carcinoma; Squamous Cell Carcinoma Metastatic in the Neck With Occult Primary; Stage IV Hypopharyngeal Squamous Cell Carcinoma; Stage IV Laryngeal Squamous Cell Carcinoma; Stage IV Laryngeal Verrucous Carcinoma; Stage IV Lip and Oral Cavity Squamous Cell Carcinoma; Stage IV Major Salivary Gland Carcinoma; Stage IV Nasal Cavity and Paranasal Sinus Squamous Cell Carcinoma; Stage IV Nasopharyngeal Keratinizing Squamous Cell Carcinoma; Stage IV Oral Cavity Verrucous Carcinoma; Stage IV Oropharyngeal Squamous Cell Carcinoma; Tongue Carcinoma; Untreated Metastatic Squamous Cell Carcinoma to Neck With Occult Primary
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Lymphoid Interstitial Pneumonia; Salivary Gland Neoplasms; Tongue Neoplasms | interventions — cediranib

ARMS (1):
- Treatment (enzyme inhibitor) (Experimental): Patients receive oral cediranib maleate once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cediranib Maleate; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Cediranib Maleate — Given orally
  Other Names: AZD2171; AZD2171 Maleate; Recentin
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well cediranib maleate works in treating patients with recurrent or newly diagnosed metastatic head and neck cancer. Cediranib maleate may stop the growth of head and neck cancer by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the objective clinical response in patients with recurrent or newly diagnosed metastatic squamous cell carcinoma of the head and neck treated with AZD2171 (cediranib maleate).

SECONDARY OBJECTIVES:

I. Determine the safety profile of this drug in these patients. II. Assess the early and late physiological and biological effects of this drug on tumor interstitial fluid pressure, pO2, and tumor microvasculature.

III. Assess the value of potential noninvasive biomarkers of response, including plasma levels of molecules involved in angiogenesis, circulating endothelial cells and progenitor cells, and functional imaging changes before and after treatment.

IV. Assess the gene expression patterns before and after treatment as predictors of clinical and biological response.

OUTLINE: This is a multicenter study.

Patients receive oral cediranib maleate once daily on days 1-28. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo dynamic contrast-enhanced CT imaging and blood collection periodically during study for research studies assessing plasma levels of angiogenic/antiangiogenic molecules, circulating endothelial cells (by flow cytometry), progenitor cells, and protein analysis of potential biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma of the head and neck meeting one of the following criteria:

  * Recurrent disease

    * Previously treated with standard curative therapy, including surgery and/or radiotherapy with or without chemotherapy
  * Newly diagnosed metastatic disease
* Must be deemed incurable by all of the following:

  * Salvage surgery
  * Radiotherapy
* Measurable disease ≥ 1 cm by conventional techniques, flexible fiberoptic laryngoscopy, or examination under anesthesia
* No more than 2 prior conventional or investigational systemic therapies for categorically incurable local-regional or distant disease
* No known primary brain tumor or brain metastases
* ECOG performance status 0-1
* Life expectancy ≥ 6 months
* WBC > 3,000/mm³
* Absolute neutrophil count > 1,500/mm³
* Platelet count > 100,000/mm³
* Hemoglobin > 8 g/dL
* Bilirubin normal
* AST and ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance > 60 mL/min
* Proteinuria ≤ +1 on 2 consecutive urine dipsticks taken ≥ 1 week apart
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* History of nonmelanoma skin cancer or other prior malignancy allowed provided the cancer has been in remission for > 3 years
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to AZD2171
* No hypertension (i.e., systolic blood pressure (BP) > 160 mm Hg and diastolic BP > 100 mm Hg)
* No history of hypertensive urgency, hypertensive emergency, or end-organ damage (i.e., thrombotic stroke, transient ischemic attacks, intracerebral hemorrhage, myocardial infarction, aortic aneurysm, or aortic dissection)
* QTc ≤ 500 msec (with Bazett's correction)
* No history of familial long QT syndrome
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Bleeding diathesis
  * Congestive heart failure, defined as New York Heart Association (NYHA) class III-IV congestive heart failure

    * NYHA class II congestive heart failure allowed provided there is increased monitoring
  * Significant ECG abnormality
  * Peripheral vascular disease
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Pulmonary edema
  * Atrioventricular (AV) conduction abnormalities
  * Sick sinus syndrome
  * Second- or third-degree AV block
  * Deep venous thrombosis
* No nonhealing ulcers, bone fracture, or wounds
* No psychiatric illness or social situation that would preclude study compliance
* No traumatic injury within the past 7 days
* No known coagulopathy that increases risk of bleeding
* No history of clinically significant hemorrhages
* See Disease Characteristics
* Recovered from all prior therapies
* No prior antiangiogenic therapy
* No more than 2 prior chemotherapy or antineoplastic regimens for categorically incurable local-regional or distant disease
* At least 4 weeks since prior radiotherapy or major surgery
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C)
* More than 30 days since prior participation in an investigational trial
* No other concurrent investigational agents
* No concurrent drugs or biologics with proarrhythmic potential
* No concurrent anticoagulants (e.g., warfarin) or antiplatelet agents
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent anticancer agents or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-02; Primary Completion 2013-05 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Tumor response (complete response [CR], partial response [PR], progressive disease [PD], and stable disease [SD]) as determined by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria | Baseline to day 29
  Compared using logistic regression.

SECONDARY OUTCOMES:
Adverse events, graded according to the revised National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | Up to 28 days after last dose of study treatment
  Analyzed using binomial confidence intervals for these proportions.
Distant metastasis | Every 2 courses until progression
  Analyzed with binomial confidence intervals as well as Kaplan-Meier estimates for these proportions.
Overall survival | Up to 28 days after last dose of study treatment
  Analyzed with binomial confidence intervals as well as Kaplan-Meier estimates for these proportions.
Progression-free survival | Up to 28 days after last dose of study treatment
  Analyzed with binomial confidence intervals as well as Kaplan-Meier estimates for these proportions.

CONTACTS AND LOCATIONS:
Overall Officials: James Rocco, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital Cancer Center, Boston, Massachusetts, United States